CLINICAL TRIAL: NCT02679859
Title: A Prospective, Multi-centre, Randomised Trial of B-type Natriuretic Peptide Guided Therapy to Improve Clinical Outcomes for Patients Undergoing Non-cardiac Surgery: the BETTER Surgery Pilot Trial
Brief Title: B-type Natriuretic Peptide Guided Therapy to Improve Clinical Outcomes for Patients Undergoing Non-cardiac Surgery
Acronym: BETTER pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of KwaZulu (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Head of Perioperative Medicine, University of Cape Town
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: No Unique ID yet
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Surgery; Cardiovascular Complications; Risk Assessment
Keywords: Natriuretic Peptide, Brain; Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B-type natriuretic guided medical therapy optimisation (Experimental): B-type natriuretic guided medical therapy optimisation
  Interventions: Other: BNP guided medical therapy optimisation
- Normal medical management (No Intervention)

INTERVENTIONS:
Other: BNP guided medical therapy optimisation
  Arms: B-type natriuretic guided medical therapy optimisation

SUMMARY:
The primary hypothesis of the BETTER pilot trial is that B-type natriuretic peptide (BNP) directed medical therapy prior to noncardiac surgery will be associated with improved cardiovascular outcomes, when compared to standard of care.

DETAILED DESCRIPTION:
Study hypothesis and aim. The primary hypothesis of the BETTER Surgery Pilot Trial is that BNP directed medical therapy prior to noncardiac surgery will be associated with improved cardiovascular outcomes, when compared to standard of care. The aim of this pilot trial is to test the feasibility of a preoperative BNP directed medical therapy trial, with the intention of then going onto a large international multicentred RCT.

Primary outcome measure. A composite of 30 day mortality, nonfatal myocardial infarction, nonfatal cardiac arrest, congestive cardiac failure and re-operation.

Secondary outcome measures.

Difference in BNP levels at the time of surgery An analysis of outcomes as a measure of achieved value i.e. the value measured immediately prior to surgery.

Duration of hospital stay Admission to critical care Time to surgery Reoperation

Trial design. A prospective, multi-centre, randomised trial of BNP guided therapy to improve clinical outcomes for patients undergoing non-cardiac surgery.

Inclusion criteria. High risk elective preoperative noncardiac surgical patients who are referred to a preanaesthetic clinic for preoperative risk stratification.

Exclusion criteria.

Patient refusal to participate Where clinical opinion suggests that surgery cannot be postponed for at least 3 to 4 weeks to allow for clinical response to a change in medical therapy Randomisation. Patients will only be randomized during the outpatient clinic visit once a decision has been taken that surgery is necessary. This will follow informed consent. Patients would be randomized to standard of care or BNP directed care. Following randomization, BNP will be measured in all patients.

1. Standard-of-care arm. These patients will be managed as per standard preoperative stratification strategies at the participating units. All personnel will be blinded to the BNP results. Optimisation of medical therapies will be encouraged.
2. BNP guided therapy patients. Based on an individual patient data meta-analysis of noncardiac surgical patients, the thresholds associated with BNP and MACE are known.

Based on these BNP thresholds, the following recommendations are made;

High risk: Additional medical therapy and/or uptitration of current therapies is strongly recommended. It is strongly recommended that surgery is deferred until the BNP falls below the high risk threshold if possible to allow for therapy response.

Intemediate risk: Additional therapy and/or uptitration of current therapies is recommended. It is recommended that surgery is deferred if possible to allow for therapy response.

Low risk: Surgery is recommended as soon as any other perioperative considerations have been addressed. Ideally, surgery is recommended at the earliest convenience.

Additional visits may also be scheduled at the discretion of the investigator for further BNP risk stratification prior to surgery at the discretion of the treating physician. Neither the attending physicians, nor the patient will be blinded to the BNP result in the BNP guided therapy arm.

BNP levels will be repeated in all patients before scheduled surgery. These preoperative BNP results will be blinded.

Irrespective of the treatment group to which the noncardiac patient has been randomized, it is recommended that all these surgical patients receive statin therapy during the perioperative period and if on aspirin, that it is stopped 72 hours before surgery, and re-instituted at 7 days postoperatively. Intraoperative and postoperative management will be at the discretion of the local physicians.

Drug therapies. Drug therapies used in the BETTER trial will be compliant with practice guidelines for heart failure therapy, up to the point of ensuring ACE-inhibition, beta-blockade and mineralocorticoid receptor antagonism. Uptitration of drugs known to decrease mortality associated with cardiac failure and secondary prevention for myocardial infarction will be considered. The minimum and maximum doses advocated in the PROTECT study have been adopted for the BETTER Surgery Pilot Trial. Uptitration will only considered where uptitration of therapy has been associated with improved survival in heart failure studies.

End point adjudication. All end points will be adjudicated by physicians blinded to treatment allocation.

Withdrawal rules. Subjects are free to voluntarily withdraw from the BETTER Surgery Trial at any time. However, events experienced by any withdrawn patient will be analyzed at the end of the trial as a function of treatment allocation under intent-to-treat considerations.

Ethics approval. Ethics approval will be obtained from each university centre. Steering committee members will ensure ethics approval is obtained from their respective centres prior to trial participation.

Data collection and collation. Access to the electronic data entry system will be protected by username and password. Username and password will be delivered during the registration process for individual local investigators. All electronic data transfer between participating centres and the co-ordinating centre will be username and password protected. Each centre will maintain a trial file including a protocol, local investigator delegation log, ethics approval documentation etc. Pseudo-anonymised (coded) data may also be sent by mail to the coordinating centre if necessary for event adjudication.

Statistical analysis. Categorical variables will be described as proportions and will be compared using chi-square or Fisher's exact test. Continuous variable will be described as mean and standard deviation if normally distributed or median and inter-quartile range if not normally distributed. Comparisons of continuous variables will be performed using one-way ANOVA or Mann-Whitney test as appropriate.

Primary clinical end point. Kaplan-Meier curves will be constructed to evaluate time to first event and compared using the log-rank test. Lastly, univariable followed by multivariable analyses will identify independent predictors of outcomes, with subsequent regression analysis performed to compare event rates, adjusting for differences between baseline variables.

It is expected that patients in the BNP guided therapy arm may end up with more repeat visits compared to the standard of care arm of the trial. To understand whether such increased contact itself is associated with better outcomes rather than a lowering of BNP, a covariate analysis controlled for total visits versus visits triggered by BNP evaluation for further therapeutic intervention, will be performed to determine the potential effect of increased visits on patient outcomes.

Trial management. Participating centres need to routinely provide preoperative risk stratification services for high risk noncardiac surgical patients. The pilot trial will be led by Bruce Biccard. Site leaders, have been identified as co-participants in this application.

Sample size calculation. For the proposed composite outcome we expect at least a 10% event rate. In a large international multicentre trial, assuming a 25% relative risk reduction in the primary outcome in the BNP directed therapy group with an event rate of 10%, we estimated a sample size of 2075 patients per group would provide a 80% power (α =0.05).

For the pilot trial we will recruit 100 patients.

How this trial will lead to a larger study.

A review of all the literature on preoperative BNP risk stratification suggests that integrating preoperative BNP into risk stratification models has reached the 4th stage integrating a biomarker into clinical practice (clinical utility). This surpasses the current Revised Cardiac Risk Index (RCRI) clinical standard in preoperative risk stratification in the process. There is good individual patient data meta-analyses which have been used to establish the BNP thresholds associated with adverse outcomes. This stresses the importance (yet lack) of randomised controlled trials which address the utility of biomarker risk stratification to improve patient outcomes through biomarker directed therapy, management and monitoring in noncardiac surgical patients. The fifth stage of integration of a biomarker into clinical practice demands demonstration that biomarker directed therapy improves clinical outcomes. A single study has been conducted in the non-surgical population, which showed a more aggressive heart failure therapy regimen driven by targetting BNP was generally well tolerated in the elderly and associated with significantly fewer cardiovascular events.

This pilot trial will assess the feasibility of such an important preoperative surgical clinical RCT. These data will be used to plan and conduct a large, multicentre RCT to address this question.

References.

1. Hlatky MA, et al. Criteria for evaluation of novel markers of cardiovascular risk: a scientific statement from the American Heart Association. Circulation. 2009;119:2408-16.
2. Biccard BM, Devereaux PJ and Rodseth RN. Cardiac biomarkers in the prediction of risk in the non-cardiac surgery setting. Anaesthesia. 2014;69:484-93.
3. Gaggin HK, et al. Heart failure outcomes and benefits of NT-proBNP-guided management in the elderly: results from the prospective, randomized ProBNP outpatient tailored chronic heart failure therapy (PROTECT) study. J Card Fail 2012;18(8):626-34.

ELIGIBILITY:
Inclusion Criteria:

* High risk elective preoperative noncardiac surgical patients who are referred to a preanaesthetic clinic for preoperative risk stratification.

Exclusion Criteria:

1. Patient refusal to participate
2. Where clinical opinion suggests that surgery cannot be postponed for at least 3 to 4 weeks to allow for clinical response to a change in medical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
A composite of 30 day mortality, nonfatal myocardial infarction, nonfatal cardiac arrest, congestive cardiac failure and re-operation. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Biccard, MD, PhD, Principal Investigator — University of Cape Town

IPD SHARING:
Plan to Share IPD: Undecided